CLINICAL TRIAL: NCT04810624
Title: Optimizing Relapse Prevention and Changing Habits in Anorexia Nervosa
Brief Title: Relapse Prevention and Changing Habits in Anorexia Nervosa
Acronym: REACH+
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: U.S. Department of Health and Human Services OHRP issued an FWA restriction on NYSPI research that included a pause of human subjects research as of June 23, 2023. This study will resume recruitment after OHRP has approved the resumption of research.
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: Columbia University (Other); Brown University (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Joanna Steinglass, Professor of Psychiatry, New York State Psychiatric Institute
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 8110; R34MH127180 (NIH)
Record Dates: First submitted 2021-01-21; First posted 2021-03-23 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-03

CONDITIONS: Anorexia Nervosa
MeSH Terms: conditions — Anorexia Nervosa | interventions — Secondary Prevention

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (26):
- Do, Accept, Motivation Through Values, Sessions, Long-Term Food Logs, (Experimental): Behavior Do: Including in-session eating experiments.
  Thought Accept: Mindfully accepting of unhelpful thoughts as passing mental phenomena that need not guide behavior.
  Motivation Through Values: Identifying individual motivators for recovery and opportunities to expand upon non-eating disorder aspects of identity.
  Sessions for Skills Consolidation: Consolidation of skills introduced to patient and monitoring of continued progress using 45-min, face-to-face (via video) sessions.
  Food Monitoring - Long-Term: Use of food logs for duration of treatment.
- Do, Accept, Motivation through Values, Sessions, Short-Term Food Logs (Experimental): Behavior Do: Including in-session eating experiments.
  Thought Accept: Mindfully accepting of unhelpful thoughts as passing mental phenomena that need not guide behavior.
  Motivation Through Values: Identifying individual motivators for recovery and opportunities to expand upon non-eating disorder aspects of identity.
  Sessions for Skills Consolidation: Consolidation of skills introduced to patient and monitoring of continued progress using 45-min, face-to-face (via video) sessions.
  Food-Monitoring - Short-Term: Use of food logs for first 5 weeks of treatment.
  Interventions: Behavioral: Relapse Prevention and Changing Habits (REACH+)
- Do, Accept, Motivation through Values, Check-Ins, Short-Term Food Logs (Experimental): Behavior Do: Including in-session eating experiments.
  Thought Accept: Mindfully accepting of unhelpful thoughts as passing mental phenomena that need not guide behavior.
  Motivation Through Values: Identifying individual motivators for recovery and opportunities to expand upon non-eating disorder aspects of identity.
  Check-Ins for Skills Consolidation: Consolidation of skills introduced to patient and monitoring of continued progress conducted independently by participant, with only brief (~20-min) check-ins during this period.
  Food-Monitoring - Short-Term: Use of food logs for first 5 weeks of treatment.
  Interventions: Behavioral: Relapse Prevention and Changing Habits (REACH+)
- Do, Accept, Motivation through Values, Check-Ins, No Food Logs (Experimental): Behavior Do: Including in-session eating experiments.
  Thought Accept: Mindfully accepting of unhelpful thoughts as passing mental phenomena that need not guide behavior.
  Motivation Through Values: Identifying individual motivators for recovery and opportunities to expand upon non-eating disorder aspects of identity.
  Check-Ins for Skills Consolidation: Consolidation of skills introduced to patient and monitoring of continued progress conducted independently by participant, with only brief (~20-min) check-ins during this period.
  No Food-Monitoring: No recommendation for food records or logs during treatment.
  Interventions: Behavioral: Relapse Prevention and Changing Habits (REACH+)
- Do, Accept, Motivation through Narratives, Sessions, Short-Term Food Logs (Experimental): Behavior Do: Including in-session eating experiments.
  Thought Accept: Mindfully accepting of unhelpful thoughts as passing mental phenomena that need not guide behavior.
  Motivation Through Narratives: Using stories of others with lived experience (e.g., writings, podcasts) to appreciate long-term dangers of AN and the opportunity for symptom resolution with sustained recovery, without discussion of individualized motivators.
  Sessions for Skills Consolidation: Consolidation of skills introduced to patient and monitoring of continued progress using 45-min, face-to-face (via video) sessions.
  Food-Monitoring - Short-Term: Use of food logs for first 5 weeks of treatment.
  Interventions: Behavioral: Relapse Prevention and Changing Habits (REACH+)
- Do, Accept, Motivation through Narratives, Sessions, No Food Logs (Experimental): Behavior Do: Including in-session eating experiments.
  Thought Accept: Mindfully accepting of unhelpful thoughts as passing mental phenomena that need not guide behavior.
  Motivation Through Narratives: Using stories of others with lived experience (e.g., writings, podcasts) to appreciate long-term dangers of AN and the opportunity for symptom resolution with sustained recovery, without discussion of individualized motivators.
  Sessions for Skills Consolidation: Consolidation of skills introduced to patient and monitoring of continued progress using 45-min, face-to-face (via video) sessions.
  No Food-Monitoring: No recommendation for food records or logs during treatment.
  Interventions: Behavioral: Relapse Prevention and Changing Habits (REACH+)
- Do, Accept, Motivation through Narratives, Check-Ins, Long-Term Food Logs (Experimental): Behavior Do: Including in-session eating experiments.
  Thought Accept: Mindfully accepting of unhelpful thoughts as passing mental phenomena that need not guide behavior.
  Motivation Through Narratives: Using stories of others with lived experience (e.g., writings, podcasts) to appreciate long-term dangers of AN and the opportunity for symptom resolution with sustained recovery, without discussion of individualized motivators.
  Check-Ins for Skills Consolidation: Consolidation of skills introduced to patient and monitoring of continued progress conducted independently by participant, with only brief (~20-min) check-ins during this period.
  Food Monitoring - Long-Term: Use of food logs for duration of treatment.
  Interventions: Behavioral: Relapse Prevention and Changing Habits (REACH+)
- Do, Change, Motivation Through Values, Sessions, Short-Term Food Logs (Experimental): Behavior Do: Including in-session eating experiments.
  Thought Change: Monitoring and actively challenging distorted thoughts.
  Motivation Through Values: Identifying individual motivators for recovery and opportunities to expand upon non-eating disorder aspects of identity.
  Sessions for Skills Consolidation: Consolidation of skills introduced to patient and monitoring of continued progress using 45-min, face-to-face (via video) sessions.
  Food-Monitoring - Short-Term: Use of food logs for first 5 weeks of treatment.
  Interventions: Behavioral: Relapse Prevention and Changing Habits (REACH+)
- Do, Change, Motivation Through Values, Sessions, No Food Logs (Experimental): Behavior Do: Including in-session eating experiments.
  Thought Change: Monitoring and actively challenging distorted thoughts.
  Motivation Through Values: Identifying individual motivators for recovery and opportunities to expand upon non-eating disorder aspects of identity.
  Sessions for Skills Consolidation: Consolidation of skills introduced to patient and monitoring of continued progress using 45-min, face-to-face (via video) sessions.
  No Food-Monitoring: No recommendation for food records or logs during treatment.
  Interventions: Behavioral: Relapse Prevention and Changing Habits (REACH+)
- Do, Change, Motivation through Values, Check-Ins, Long-Term Food Logs (Experimental): Behavior Do: Including in-session eating experiments.
  Thought Change: Monitoring and actively challenging distorted thoughts.
  Motivation Through Values: Identifying individual motivators for recovery and opportunities to expand upon non-eating disorder aspects of identity.
  Check-Ins for Skills Consolidation: Consolidation of skills introduced to patient and monitoring of continued progress conducted independently by participant, with only brief (~20-min) check-ins during this period.
  Food Monitoring - Long-Term: Use of food logs for duration of treatment.
  Interventions: Behavioral: Relapse Prevention and Changing Habits (REACH+)
- Do, Change, Motivation Through Narratives, Sessions, Long-term Food Logs (Experimental): Behavior Do: Including in-session eating experiments.
  Thought Change: Monitoring and actively challenging distorted thoughts.
  Motivation Through Narratives: Using stories of others with lived experience (e.g., writings, podcasts) to appreciate long-term dangers of AN and the opportunity for symptom resolution with sustained recovery, without discussion of individualized motivators.
  Sessions for Skills Consolidation: Consolidation of skills introduced to patient and monitoring of continued progress using 45-min, face-to-face (via video) sessions.
  Food Monitoring - Long-Term: Use of food logs for duration of treatment.
  Interventions: Behavioral: Relapse Prevention and Changing Habits (REACH+)
- Talk, Accept, Motivation through Values, Sessions, Short-Term Food Logs (Experimental): Behavior Talk: Discussion of recent eating and plans for upcoming eating; absence of in-session eating experiments.
  Thought Accept: Mindfully accepting of unhelpful thoughts as passing mental phenomena that need not guide behavior.
  Motivation Through Values: Identifying individual motivators for recovery and opportunities to expand upon non-eating disorder aspects of identity.
  Sessions for Skills Consolidation: Consolidation of skills introduced to patient and monitoring of continued progress using 45-min, face-to-face (via video) sessions.
  Food-Monitoring - Short-Term: Use of food logs for first 5 weeks of treatment.
  Interventions: Behavioral: Relapse Prevention and Changing Habits (REACH+)
- Talk, Accept, Motivation through Values, Sessions, No Food Logs (Experimental): Behavior Talk: Discussion of recent eating and plans for upcoming eating; absence of in-session eating experiments.
  Thought Accept: Mindfully accepting of unhelpful thoughts as passing mental phenomena that need not guide behavior.
  Motivation Through Values: Identifying individual motivators for recovery and opportunities to expand upon non-eating disorder aspects of identity.
  Sessions for Skills Consolidation: Consolidation of skills introduced to patient and monitoring of continued progress using 45-min, face-to-face (via video) sessions.
  No Food-Monitoring: No recommendation for food records or logs during treatment.
  Interventions: Behavioral: Relapse Prevention and Changing Habits (REACH+)
- Talk, Accept, Motivation through Narratives, Check-Ins, Short-Term Food Logs (Experimental): Behavior Talk: Discussion of recent eating and plans for upcoming eating; absence of in-session eating experiments.
  Thought Accept: Mindfully accepting of unhelpful thoughts as passing mental phenomena that need not guide behavior.
  Motivation Through Narratives: Using stories of others with lived experience (e.g., writings, podcasts) to appreciate long-term dangers of AN and the opportunity for symptom resolution with sustained recovery, without discussion of individualized motivators.
  Check-Ins for Skills Consolidation: Consolidation of skills introduced to patient and monitoring of continued progress conducted independently by participant, with only brief (~20-min) check-ins during this period.
  Food-Monitoring - Short-Term: Use of food logs for first 5 weeks of treatment.
  Interventions: Behavioral: Relapse Prevention and Changing Habits (REACH+)
- Talk, Accept, Motivation through Narratives, Check-Ins, No Food Logs (Experimental): Behavior Talk: Discussion of recent eating and plans for upcoming eating; absence of in-session eating experiments.
  Thought Accept: Mindfully accepting of unhelpful thoughts as passing mental phenomena that need not guide behavior.
  Motivation Through Narratives: Using stories of others with lived experience (e.g., writings, podcasts) to appreciate long-term dangers of AN and the opportunity for symptom resolution with sustained recovery, without discussion of individualized motivators.
  Check-Ins for Skills Consolidation: Consolidation of skills introduced to patient and monitoring of continued progress conducted independently by participant, with only brief (~20-min) check-ins during this period.
  No Food-Monitoring: No recommendation for food records or logs during treatment.
  Interventions: Behavioral: Relapse Prevention and Changing Habits (REACH+)
- Talk, Change, Motivation Through Values, Sessions, Long-Term Food Logs (Experimental): Behavior Talk: Discussion of recent eating and plans for upcoming eating; absence of in-session eating experiments.
  Thought Change: Monitoring and actively challenging distorted thoughts.
  Motivation Through Values: Identifying individual motivators for recovery and opportunities to expand upon non-eating disorder aspects of identity.
  Sessions for Skills Consolidation: Consolidation of skills introduced to patient and monitoring of continued progress using 45-min, face-to-face (via video) sessions.
  Food Monitoring - Long-Term: Use of food logs for duration of treatment.
  Interventions: Behavioral: Relapse Prevention and Changing Habits (REACH+)
- Talk, Change, Motivation Through Values, Sessions, No Food Logs (Experimental): Behavior Talk: Discussion of recent eating and plans for upcoming eating; absence of in-session eating experiments.
  Thought Change: Monitoring and actively challenging distorted thoughts.
  Motivation Through Values: Identifying individual motivators for recovery and opportunities to expand upon non-eating disorder aspects of identity.
  Sessions for Skills Consolidation: Consolidation of skills introduced to patient and monitoring of continued progress using 45-min, face-to-face (via video) sessions.
  No Food-Monitoring: No recommendation for food records or logs during treatment.
  Interventions: Behavioral: Relapse Prevention and Changing Habits (REACH+)
- Talk, Change, Motivation through Values, Check-Ins, Short-Term Food Logs (Experimental): Behavior Talk: Discussion of recent eating and plans for upcoming eating; absence of in-session eating experiments.
  Thought Change: Monitoring and actively challenging distorted thoughts.
  Motivation Through Values: Identifying individual motivators for recovery and opportunities to expand upon non-eating disorder aspects of identity.
  Check-Ins for Skills Consolidation: Consolidation of skills introduced to patient and monitoring of continued progress conducted independently by participant, with only brief (~20-min) check-ins during this period.
  Food-Monitoring - Short-Term: Use of food logs for first 5 weeks of treatment.
  Interventions: Behavioral: Relapse Prevention and Changing Habits (REACH+)
- Talk, Change, Motivation through Values, Check-Ins, No Food Logs (Experimental): Behavior Talk: Discussion of recent eating and plans for upcoming eating; absence of in-session eating experiments.
  Thought Change: Monitoring and actively challenging distorted thoughts.
  Motivation Through Values: Identifying individual motivators for recovery and opportunities to expand upon non-eating disorder aspects of identity.
  Check-Ins for Skills Consolidation: Consolidation of skills introduced to patient and monitoring of continued progress conducted independently by participant, with only brief (~20-min) check-ins during this period.
  No Food-Monitoring: No recommendation for food records or logs during treatment.
  Interventions: Behavioral: Relapse Prevention and Changing Habits (REACH+)
- Talk, Change, Motivation through Narratives, Sessions, Short-Term Food Logs (Experimental): Behavior Talk: Discussion of recent eating and plans for upcoming eating; absence of in-session eating experiments.
  Thought Change: Monitoring and actively challenging distorted thoughts.
  Motivation Through Narratives: Using stories of others with lived experience (e.g., writings, podcasts) to appreciate long-term dangers of AN and the opportunity for symptom resolution with sustained recovery, without discussion of individualized motivators.
  Sessions for Skills Consolidation: Consolidation of skills introduced to patient and monitoring of continued progress using 45-min, face-to-face (via video) sessions.
  Food-Monitoring - Short-Term: Use of food logs for first 5 weeks of treatment.
  Interventions: Behavioral: Relapse Prevention and Changing Habits (REACH+)
- Talk, Change, Motivation through Narratives, Sessions, No Food Logs (Experimental): Behavior Talk: Discussion of recent eating and plans for upcoming eating; absence of in-session eating experiments.
  Thought Change: Monitoring and actively challenging distorted thoughts.
  Motivation Through Narratives: Using stories of others with lived experience (e.g., writings, podcasts) to appreciate long-term dangers of AN and the opportunity for symptom resolution with sustained recovery, without discussion of individualized motivators.
  Sessions for Skills Consolidation: Consolidation of skills introduced to patient and monitoring of continued progress using 45-min, face-to-face (via video) sessions.
  No Food-Monitoring: No recommendation for food records or logs during treatment.
  Interventions: Behavioral: Relapse Prevention and Changing Habits (REACH+)
- Talk, Change, Motivation through Narratives, Check-Ins, Long-Term Food Logs (Experimental): Behavior Talk: Discussion of recent eating and plans for upcoming eating; absence of in-session eating experiments.
  Thought Change: Monitoring and actively challenging distorted thoughts.
  Motivation Through Narratives: Using stories of others with lived experience (e.g., writings, podcasts) to appreciate long-term dangers of AN and the opportunity for symptom resolution with sustained recovery, without discussion of individualized motivators.
  Check-Ins for Skills Consolidation: Consolidation of skills introduced to patient and monitoring of continued progress conducted independently by participant, with only brief (~20-min) check-ins during this period.
  Food Monitoring - Long-Term: Use of food logs for duration of treatment.
  Interventions: Behavioral: Relapse Prevention and Changing Habits (REACH+)
- Do, Change, Motivation through Narratives, Check-Ins, Short-Term Food Logs (Experimental): Behavior Do: Including in-session eating experiments.
  Thought Change: Monitoring and actively challenging distorted thoughts.
  Motivation Through Narratives: Using stories of others with lived experience (e.g., writings, podcasts) to appreciate long-term dangers of AN and the opportunity for symptom resolution with sustained recovery, without discussion of individualized motivators.
  Check-Ins for Skills Consolidation: Consolidation of skills introduced to patient and monitoring of continued progress conducted independently by participant, with only brief (~20-min) check-ins during this period.
  Food-Monitoring - Short-Term: Use of food logs for first 5 weeks of treatment.
  Interventions: Behavioral: Relapse Prevention and Changing Habits (REACH+)
- Do, Change, Motivation through Narratives, Check-Ins, No Food Logs (Experimental): Behavior Do: Including in-session eating experiments.
  Thought Change: Monitoring and actively challenging distorted thoughts.
  Motivation Through Narratives: Using stories of others with lived experience (e.g., writings, podcasts) to appreciate long-term dangers of AN and the opportunity for symptom resolution with sustained recovery, without discussion of individualized motivators.
  Check-Ins for Skills Consolidation: Consolidation of skills introduced to patient and monitoring of continued progress conducted independently by participant, with only brief (~20-min) check-ins during this period.
  No Food-Monitoring: No recommendation for food records or logs during treatment.
  Interventions: Behavioral: Relapse Prevention and Changing Habits (REACH+)
- Talk, Accept, Motivation through Values, Check-Ins, Long-Term Food Logs (Experimental): Behavior Talk: Discussion of recent eating and plans for upcoming eating; absence of in-session eating experiments.
  Thought Accept: Mindfully accepting of unhelpful thoughts as passing mental phenomena that need not guide behavior.
  Motivation Through Values: Identifying individual motivators for recovery and opportunities to expand upon non-eating disorder aspects of identity.
  Check-Ins for Skills Consolidation: Consolidation of skills introduced to patient and monitoring of continued progress conducted independently by participant, with only brief (~20-min) check-ins during this period.
  Food Monitoring - Long-Term: Use of food logs for duration of treatment.
  Interventions: Behavioral: Relapse Prevention and Changing Habits (REACH+)
- Talk, Accept, Motivation through Narratives, Sessions, Long-Term Food Logs (Experimental): Behavior Talk: Discussion of recent eating and plans for upcoming eating; absence of in-session eating experiments.
  Thought Accept: Mindfully accepting of unhelpful thoughts as passing mental phenomena that need not guide behavior.
  Motivation Through Narratives: Using stories of others with lived experience (e.g., writings, podcasts) to appreciate long-term dangers of AN and the opportunity for symptom resolution with sustained recovery, without discussion of individualized motivators.
  Sessions for Skills Consolidation: Consolidation of skills introduced to patient and monitoring of continued progress using 45-min, face-to-face (via video) sessions.
  Food Monitoring - Long-Term: Use of food logs for duration of treatment.
  Interventions: Behavioral: Relapse Prevention and Changing Habits (REACH+)

INTERVENTIONS:
Behavioral: Relapse Prevention and Changing Habits (REACH+) — Psychotherapy
  Arms: Do, Accept, Motivation through Narratives, Check-Ins, Long-Term Food Logs; Do, Accept, Motivation through Narratives, Sessions, No Food Logs; Do, Accept, Motivation through Narratives, Sessions, Short-Term Food Logs; Do, Accept, Motivation through Values, Check-Ins, No Food Logs; Do, Accept, Motivation through Values, Check-Ins, Short-Term Food Logs; Do, Accept, Motivation through Values, Sessions, Short-Term Food Logs; Do, Change, Motivation Through Narratives, Sessions, Long-term Food Logs; Do, Change, Motivation Through Values, Sessions, No Food Logs; Do, Change, Motivation Through Values, Sessions, Short-Term Food Logs; Do, Change, Motivation through Narratives, Check-Ins, No Food Logs; Do, Change, Motivation through Narratives, Check-Ins, Short-Term Food Logs; Do, Change, Motivation through Values, Check-Ins, Long-Term Food Logs; Talk, Accept, Motivation through Narratives, Check-Ins, No Food Logs; Talk, Accept, Motivation through Narratives, Check-Ins, Short-Term Food Logs; Talk, Accept, Motivation through Narratives, Sessions, Long-Term Food Logs; Talk, Accept, Motivation through Values, Check-Ins, Long-Term Food Logs; Talk, Accept, Motivation through Values, Sessions, No Food Logs; Talk, Accept, Motivation through Values, Sessions, Short-Term Food Logs; Talk, Change, Motivation Through Values, Sessions, Long-Term Food Logs; Talk, Change, Motivation Through Values, Sessions, No Food Logs; Talk, Change, Motivation through Narratives, Check-Ins, Long-Term Food Logs; Talk, Change, Motivation through Narratives, Sessions, No Food Logs; Talk, Change, Motivation through Narratives, Sessions, Short-Term Food Logs; Talk, Change, Motivation through Values, Check-Ins, No Food Logs; Talk, Change, Motivation through Values, Check-Ins, Short-Term Food Logs

SUMMARY:
This study aims to optimize a treatment package for the relapse prevention treatment of AN. In the Preparation Phase, we examined accessibility and feasibility of the treatment package.

In the current Optimization Phase, we will identify which components of treatment contribute to positive outcomes after acute hospitalization. We will carefully evaluate maintenance of remission, measured by rate of weight loss and end-of-trial status.

DETAILED DESCRIPTION:
While many approaches to reducing relapse after hospital care have been tried, there is little information about which treatment elements confer benefit. This trial, Relapse Prevention and Changing Habits (REACH+), targets the habitual control of maladaptive behavior to support patients with AN in the 6 months after acute treatment, a time of high vulnerability to relapse. Each component of REACH+ addresses a question that is critical to answer in order to identify and optimize a relapse prevention treatment package that balances efficacy and burden. We will test the acceptability and feasibility of 5 components that together target habits: 1) Behavioral, 2) Cognitive, 3)Motivation, 4) Food Monitoring, and 5) Skill Consolidation. In the Preparation Phase, 10 participants were enrolled, and accessibility and feasibility of the treatment package was examined. The current Optimization Phase includes a finalized treatment manual (including an online platform) and will test each component's contribution to weight maintenance after acute treatment.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Anorexia Nervosa at hospital admission
* Medically Stable
* Internet capability with videoconferencing
* Weight restored (BMI > 19 kg/m2) at New York State Psychiatric Institute

Exclusion Criteria:

* Current substance use or other comorbid disorder requiring specialized treatment
* Pregnancy
* Imminent risk of suicide
* Serious medical illness
* Daily psychotropic medication other than antidepressants (medications that are known effect weight are exclusionary, i.e. stimulants, olanzapine, mirtazapine)
* Participation in outside psychotherapy or structured treatment program (support groups will be allowed). Individuals who are discharged on medications would need to have a non-study psychiatrist.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-06-21 (Actual); Primary Completion 2026-01-30 (Estimated); Study Completion 2026-01-30 (Estimated)

PRIMARY OUTCOMES:
Weight maintenance | 6-month end of treatment
  Measured via rate of weight loss (in lbs) following discharge from inpatient unit

SECONDARY OUTCOMES:
Habit strength | 6-month end of treatment
  Measured via Self-Report Habit Index (SRHI)
Weight/shape distortion | 6-month end of treatment
  Measured via Eating Disorder Examination, Questionnaire Version (EDE-Q)
Intrinsic motivation | 6-month end of treatment
  Measured via General Self-Efficacy Scale (GSES)
Dietary restriction | 6-month end of treatment
  Measured via Food Choice Task
Skill consolidation | 6-month end of treatment
  Measured via platform utilization time

CONTACTS AND LOCATIONS:
Locations (1):
- New York State Psychiatric Institute, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Steinglass JE, Attia E, Glasofer DR, Wang Y, Ruggiero J, Walsh BT, Thomas JG. Optimizing relapse prevention and changing habits (REACH+) in anorexia nervosa. Int J Eat Disord. 2022 Jun;55(6):851-857. doi: 10.1002/eat.23724. Epub 2022 Apr 30. PMID 35488866